CLINICAL TRIAL: NCT02274740
Title: Effect of GLP-1 Receptors Agonist Lixisenatide on Postprandial Lipid Profile in Obese Type 2 Diabetic Patients
Brief Title: Effect of Lixisenatide on Postprandial Lipid Profile in Obese Type 2 Diabetic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision not related to safety reasons
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIXISL07016; U1111-1153-3774 (Other: UTN)
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lixisenatide (Experimental): Lixisenatide injection should be performed in the morning, within 1 hour (ie, 0-60 minutes), prior to breakfast (or standardized meal).
  Lixisenatide is to be started with once daily injections of 10 μg per day for 2 weeks then to be continued by the maintenance dose (8 weeks) of 20 μg/d up to the end of the treatment period.
  Interventions: Drug: LIXISENATIDE AVE0010; Drug: metformin
- metformin (No Intervention): Greater than or equal than 1.5 g/day as background therapy for 10 weeks

INTERVENTIONS:
Drug: LIXISENATIDE AVE0010 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: lixisenatide
Drug: metformin — Pharmaceutical form:tablet Route of administration: oral
  Arms: lixisenatide

SUMMARY:
Primary Objective:

To evaluate the ability of lixisenatide to modulate postprandial hyperlipidemia in particular, the effects on plasma changes in triglycerides.

Secondary Objectives:

The effect of lixisenatide on the following postprandial lipids: apolipoprotein (APO) B48; free fatty acid, lipoprotein distribution, cholesterol, and low-density lipoprotein (LDL) oxidation.

The effect of lixisenatide on chronic low-grade inflammation present in non-insulin dependent diabetes mellitus (NIDDM) and obesity.

The effect of lixisenatide on microvascular dysfunction. To evaluate the effect of lixisenatide on postprandial plasma glucose, insulin and C-peptide and glucagon.

DETAILED DESCRIPTION:
Maximum study duration of approximately 2.5 months (study treatment) ± 2 days Day 0 (baseline) plus a 10-week open-label, active-controlled treatment period (Final/End-of-treatment Visit).

ELIGIBILITY:
Inclusion criteria:

Male and female patients, 18-70 years of age.

Diagnosis of Type 2 diabetes treated with metformin and obesity (body mass index [BMI] >30 kg/m^2) and the following other abnormalities:

* Abdominal obesity (waist circumference >102 cm in men and >88 cm in women). According to National Cholesterol Education Program-Adult Treatment Panel (NCEP-ATP) III (2001).
* Glycated hemoglobin A1c (HbA1c) ≥7 and ≤8.5% (after Sponsor approval providers might reasonably suggest more stringent A1c goals [such as 6.5%] for selected individual patients, if this can be achieved without significant hypoglycemia or other adverse effects of treatment. Appropriate patients might include those with short duration of diabetes, long life expectancy, and no significant cardiovascular disease).
* Hypertriglyceridemia (fasting triglyceride levels between 150 mg/dL and 600 mg/dL, cholesterol <300 mg/dL. In order to exclude patients who might be suffering from a primitive dyslipidemia).
* Low high-density lipoprotein (HDL) cholesterol (serum HDL-cholesterol <40 mg/dL in men and <50 mg/dL in women).

Written informed consent.

Exclusion criteria:

Smoking. Thyroid disease even if under appropriate hormonal replacement therapy or thyroid suppressant (Thyroid Stimulating Hormone [TSH] >5 mU/L with clinical symptoms of hypothyroidism).

Hepatic disease (Aspartate Aminotransferase [ASAT] or Alanine Aminotransferase [ALAT] >2 times the upper limit of normal).

Renal disease (serum creatinine >1.7 times the upper limit of normal). A history of coronary heart disease, cerebrovascular disease, or peripheral arterial disease in the 6 months before enrollment.

History of malignancies. Use of lipid lowering therapy. Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg. Triglycerides >600 mg/dL. History of chronic pancreatitis or of idiopathic acute pancreatitis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in plasma triglycerides after 10 weeks of treatment area under-the-time concentration curve between 0 and 480 minutes (AUC0-480 min) | After 10 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in plasma triglyceride | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in plasma cholesterol | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in APO B48 | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in free fatty acid levels | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in lipoprotein distribution | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in LDL oxidation | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in postprandial plasma glucose | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in insulin | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in C-peptide | 2 days after the basal test and after 10 weeks of treatment
Change from baseline in low grade inflammation (cytokines and stress oxidative markers) | 2 days after the basal test and after 10 weeks of treatment
Change in baseline coronary flow reserve to assess the effect of lixisenatide on microvascular dysfunction | 2 days after the basal test and after 10 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi